CLINICAL TRIAL: NCT00794625
Title: Adjunctive Treatment With Divalproex or Risperidone for Aggression Refractory to Stimulant Monotherapy Among Children With ADHD
Brief Title: Effectiveness of Combined Medication Treatment for Aggression in Children With Attention Deficit With Hyperactivity Disorder (The SPICY Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joseph Blader (NIH)
Collaborators: University of Texas (Other); Northwell Health (Other)
Responsible Party: Sponsor-Investigator, Joseph Blader, Associate Professor of Psychiatry, Stony Brook State University of New York, National Institute of Mental Health (NIMH)
Organization: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01MH080050 (NIH); DSIR 84-CTM
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention-Deficit/Hyperactivity Disorder; Aggressive Behavior; Oppositional Defiant Disorder; Conduct Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Aggression; Oppositional Defiant Disorder; Conduct Disorder | interventions — Valproic Acid; Risperidone; Sugars; Methylphenidate; Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): During Phase 1, participants will receive a stimulant medication. If they do not respond to the stimulant, they will add valproate and behavioral family counseling to their treatment during Phase 2. If they do not respond to valproate, they will be switched to risperidone.
  Interventions: Drug: Valproate; Drug: Risperidone; Drug: Stimulant medication; Behavioral: Behavioral family counseling
- 2 (Experimental): During Phase 1, participants will receive a stimulant medication. If they do not respond to the stimulant, they will add risperidone and behavioral family counseling to their treatment during Phase 2. If they do not respond to risperidone, they will switch to valproate.
  Interventions: Drug: Valproate; Drug: Risperidone; Drug: Stimulant medication; Behavioral: Behavioral family counseling
- 3 (Placebo Comparator): During Phase 1, participants will receive a stimulant medication. If they do not respond to the stimulant, they will add placebo and behavioral family counseling to their treatment during Phase 2.
  Interventions: Drug: Placebo; Drug: Stimulant medication; Behavioral: Behavioral family counseling

INTERVENTIONS:
Drug: Valproate — Standard therapeutic doses of valproate, set according to valproic acid blood level, for 8 weeks
  Other Names: Depakote; Valproic acid
  Arms: 1; 2
Drug: Risperidone — Standard therapeutic doses of risperidone for 8 weeks
  Other Names: Risperdal
  Arms: 1; 2
Drug: Placebo — An inactive substance at identical dosing to active treatments for 8 weeks
  Other Names: Inactive substance; "Sugar pill"
  Arms: 3
Drug: Stimulant medication — Stimulant medication standard in the care of ADHD, such as methylphenidate or dextroamphetamine
  Other Names: Ritalin; Dexedrine
Behavioral: Behavioral family counseling — Weekly behavioral counseling with a therapist

SUMMARY:
This study will determine the advantages and disadvantages of adding one of two different types of drugs to stimulant treatment for reducing aggressive behavior in children with attention deficit with hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
Attention deficit with hyperactivity disorder (ADHD) is a common childhood mental disorder that affects 3% to 5% of all American children. Symptoms of ADHD commonly include inability to focus or exercise normal inhibition, and in some cases, aggressive behavior. Approximately 33% to 50% of children with ADHD develop oppositional defiant disorder (ODD), and about 20% to 40% develop a conduct disorder (CD). These disorders are characterized by defiant, belligerent, and otherwise aggressive behavior. Treatment for ADHD generally includes use of stimulant medications that decrease impulsivity and increase attentiveness, such as methylphenidate (Ritalin) or dextroamphetamine (Dexedrine), but these do not always affect aggression. To treat aggression in ADHD, many physicians prescribe additional medications, including the mood stabilizing medication valproate and the antipsychotic medication risperidone.

There is no clinical evidence proving that using multiple types of medications is safe and effective. This study will treat children with ADHD and aggression with a combination of stimulants and antipsychotic or mood stabilizing medications to determine whether the aggressive behaviors and ADHD symptoms are reduced without harmful side effects.

This study has two phases. During the first phase, which will last 3 to 6 weeks, participants will be treated with normal ADHD stimulant medications. During the second phase, those whose aggressive behavior is not effectively suppressed by stimulant medication alone will then be randomly assigned to also receive valproate, risperidone, or placebo for 8 weeks. After 8 weeks, children whose aggression persists will be switched from either valproate to risperidone or risperidone to valproate for another 8 weeks. Those on placebo will not switch medications. All participants will attend weekly monitoring visits for 11 to 16 weeks over the course of the study. At these visits, aggression levels and medication side effects will be assessed. Families will also meet with the researchers to discuss the child's progress and will attend behavioral counseling with a therapist.

ELIGIBILITY:
Inclusion Criteria:

* Presence of ADHD
* Presence of persistent, clinically significant aggression
* Presence of ODD or CD

Exclusion Criteria:

* Presence of psychosis
* Presence of a major developmental disability
* Presence of a major mood disorder
* Contraindications to stimulant, valproate, or risperidone treatment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-11 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Aggressive behavior | Measured weekly for 11 to 16 weeks

SECONDARY OUTCOMES:
ADHD symptoms | Measured weekly for 11 to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C. Blader, PhD, MSc, Principal Investigator — Stony Brook University School of Medicine, State University of New York
Locations (3):
- United States (3):
  - North Shore - LIJ Health System, Zucker Hillside Hospital, Glen Oaks, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Blader JC, Pliszka SR, Kafantaris V, Foley CA, Carlson GA, Crowell JA, Bailey BY, Sauder C, Daviss WB, Sinha C, Matthews TL, Margulies DM. Stepped Treatment for Attention-Deficit/Hyperactivity Disorder and Aggressive Behavior: A Randomized, Controlled Trial of Adjunctive Risperidone, Divalproex Sodium, or Placebo After Stimulant Medication Optimization. J Am Acad Child Adolesc Psychiatry. 2021 Feb;60(2):236-251. doi: 10.1016/j.jaac.2019.12.009. Epub 2020 Jan 30. PMID 32007604
- [Derived] Blader JC, Pliszka SR, Kafantaris V, Sauder C, Posner J, Foley CA, Carlson GA, Crowell JA, Margulies DM. Prevalence and Treatment Outcomes of Persistent Negative Mood Among Children with Attention-Deficit/Hyperactivity Disorder and Aggressive Behavior. J Child Adolesc Psychopharmacol. 2016 Mar;26(2):164-73. doi: 10.1089/cap.2015.0112. Epub 2016 Jan 8. PMID 26745211
- [Derived] Blader JC, Pliszka SR, Kafantaris V, Foley CA, Crowell JA, Carlson GA, Sauder CL, Margulies DM, Sinha C, Sverd J, Matthews TL, Bailey BY, Daviss WB. Callous-unemotional traits, proactive aggression, and treatment outcomes of aggressive children with attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2013 Dec;52(12):1281-93. doi: 10.1016/j.jaac.2013.08.024. Epub 2013 Sep 25. PMID 24290461